CLINICAL TRIAL: NCT05394896
Title: Hypotension Prediction With HPI Algorithm During Decessed-donor Kidney Transplant: an Explorative, Monocentric, RCT
Brief Title: Hypotension Prediction With HPI Algorithm During Decessed-donor Kidney Transplant (HPI2022)
Acronym: HPI2022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Cristiana Laici, MD, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPI2022
Record Dates: First submitted 2022-05-22; First posted 2022-05-27 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hypotension During Surgery; Kidney Transplant; Complications
Keywords: HPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI group (Experimental): Conventional therapy and monitoring with ACUMEN sensor (Edwards Lifesciences, Irvine, USA) and Hemosphere platform (Edwards Lifesciences, Irvine, USA) of invasive blood pressure. Strategy to prevent hypotension based on HPI index, Eadyn and dP/dTmax.
  Interventions: Device: ACUMEN (Edwards Lifesciences, Irvine, USA)
- Control group (Active Comparator): Conventional therapy according to standard monitoring in the operating room which includes invasive blood pressure monitoring.
  Interventions: Device: Invasive Blood Pressure

INTERVENTIONS:
Device: ACUMEN (Edwards Lifesciences, Irvine, USA) — ACUMEN sensor generates HPI index which should predict hypotension. Based on HPI index, Eadyn and dP/dTmax values anaesthesia should somministrate liquid or drugs to prevent hypotension.
  Arms: HPI group
Device: Invasive Blood Pressure — Invasive Blood Pressure permits continue monitoring of blood pressure (routine standard for kidney transplant surgery)
  Arms: Control group

SUMMARY:
HPI monitoring and the adoption of therapeutic interventions before hypotension occurs should be ensure a shorter time of intra-operative hypotension (MAP < 65 mmHg) during deceased-donor kidney transplant surgery. The control group is represented by patients undergoing the same surgical procedure with hemodynamic monitoring with invasive blood pressure monitoring which represents the gold standard for this surgery. HPI monitoring has not yet been investigated during this surgery.

ELIGIBILITY:
Inclusion Criteria:

* First single or double kidney transplant from a cadaveric donor;
* ASA Class III-IV;
* Signature of informed consent.

Exclusion Criteria:

* Patient with atrial fibrillation rhythm or high frequency tachyarrhythmias;
* Severe valvulopathies;
* Combined single/double kidney-liver-transplant;
* Patients in whom the need for monitoring would still be expected advanced, invasive or minimally invasive hemodynamic, regardless of the allocation to the study group;
* Inclusion in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Intra-operative hypotension time | From 20 minutes after anaesthesia induction to the end of surgery (intra-operative)
  Hypotension (MAP < 65 mmHg) time relative to the range from 20 minutes after induction to the end of surgery

SECONDARY OUTCOMES:
Post-operative hypotension time | From the end of surgery to the first 12 hours after surgery (post-operative)
  Hypotension (MAP < 65 mmHg) time relative to the range from the end of surgery to the first 12 hours after surgery
Intra-operative severe hypotension time | From 20 minutes after anaesthesia induction to the end of surgery (intra-operative)
  Severe hypotension (MAP < 50 mmHg) time relative to the range from 20 minutes after induction to the end of surgery
Major Adverse Cardiovascular Events (MACE) | First 5 post-operative days after surgery (post-operative)
  Number of major cardiovascular complications (MACE) within the first five days after kidney transplantation (for MACE the composite endpoint of heart attack is considered heart failure, heart failure or presumed cardiac death)
Hospital mortality | First 30 post-operative days after surgery (post-operative)
  Number of patient died in the first 30 days after surgery
Intensive Care Unit Length of Stay | First 30 post-operative days after surgery (post-operative)
  Number of hours of ICU admission
Hospital Length of Stay | First 30 post-operative days after surgery (post-operative)
  Number of days before hospital discharge
Delayed Graft Function (DGF) | First 7 post-operative days (post-operative)
  Need for hemodialysis in first 7 postoperative days
Graft survival | 30 days after transplantation
Post-operative delirium | First 5 post-operative days
  CAM-ICU positive (asses one time for a day in the first 5 postoperative days)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biancofiore G, Cecconi M, Rocca GD. A web-based Italian survey of current trends, habits and beliefs in hemodynamic monitoring and management. J Clin Monit Comput. 2015 Oct;29(5):635-42. doi: 10.1007/s10877-014-9646-7. Epub 2014 Dec 12. PMID 25500761
- [Background] Perilli V, Aceto P, Sacco T, Modesti C, Ciocchetti P, Vitale F, Russo A, Fasano G, Dottorelli A, Sollazzi L. Anaesthesiological strategies to improve outcome in liver transplantation recipients. Eur Rev Med Pharmacol Sci. 2016 Jul;20(15):3172-7. PMID 27466988
- [Background] Vincent JL, Rhodes A, Perel A, Martin GS, Della Rocca G, Vallet B, Pinsky MR, Hofer CK, Teboul JL, de Boode WP, Scolletta S, Vieillard-Baron A, De Backer D, Walley KR, Maggiorini M, Singer M. Clinical review: Update on hemodynamic monitoring--a consensus of 16. Crit Care. 2011 Aug 18;15(4):229. doi: 10.1186/cc10291. PMID 21884645
- [Background] Lobo SM, Rezende E, Knibel MF, Silva NB, Paramo JA, Nacul FE, Mendes CL, Assuncao M, Costa RC, Grion CC, Pinto SF, Mello PM, Maia MO, Duarte PA, Gutierrez F, Silva JM Jr, Lopes MR, Cordeiro JA, Mellot C. Early determinants of death due to multiple organ failure after noncardiac surgery in high-risk patients. Anesth Analg. 2011 Apr;112(4):877-83. doi: 10.1213/ANE.0b013e3181e2bf8e. Epub 2010 Jun 8. PMID 20530615
- [Background] Pearse RM, Harrison DA, James P, Watson D, Hinds C, Rhodes A, Grounds RM, Bennett ED. Identification and characterisation of the high-risk surgical population in the United Kingdom. Crit Care. 2006;10(3):R81. doi: 10.1186/cc4928. Epub 2006 Jun 2. PMID 16749940
- [Background] Jhanji S, Thomas B, Ely A, Watson D, Hinds CJ, Pearse RM. Mortality and utilisation of critical care resources amongst high-risk surgical patients in a large NHS trust. Anaesthesia. 2008 Jul;63(7):695-700. doi: 10.1111/j.1365-2044.2008.05560.x. Epub 2008 May 16. PMID 18489613
- [Background] Fischer MO, Fiant AL, Boutros M, Flais F, Filipov T, Debroczi S, Pasqualini L, Rhanem T, Gerard JL, Guittet L, Hanouz JL, Alves A, Parienti JJ; PANEX3 study group. Perioperative hemodynamic optimization using the photoplethysmography in colorectal surgery (the PANEX3 trial): study protocol for a randomized controlled trial. Trials. 2016 Mar 22;17:159. doi: 10.1186/s13063-016-1278-4. PMID 27004412
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Background] Gomez-Izquierdo JC, Feldman LS, Carli F, Baldini G. Meta-analysis of the effect of goal-directed therapy on bowel function after abdominal surgery. Br J Surg. 2015 May;102(6):577-89. doi: 10.1002/bjs.9747. Epub 2015 Mar 11. PMID 25759947
- [Background] Walsh SR, Tang T, Bass S, Gaunt ME. Doppler-guided intra-operative fluid management during major abdominal surgery: systematic review and meta-analysis. Int J Clin Pract. 2008 Mar;62(3):466-70. doi: 10.1111/j.1742-1241.2007.01516.x. Epub 2007 Nov 21. PMID 18031528